CLINICAL TRIAL: NCT03853070
Title: Post Market Clinical Follow-Up for ED Coil / Electro-detach Generator v4
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaneka Corporation (Industry)
Collaborators: ClinSearch (Other)
Responsible Party: Sponsor
Other Study IDs: ED Coil Prosp
Record Dates: First submitted 2019-02-11; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Aneurysm; Arteriovenous Malformations; Arterio-venous Fistula
MeSH Terms: conditions — Aneurysm; Arteriovenous Malformations; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ED Coil / Electro-detach Generator v4 — The ED Coil is used for vascular embolization with a platinum coil at the target lesion in a patient's blood vessel. The ED Detach Generator is intended to for use solely to detach the platinum coil from the delivery catheter of the ED Coil.

SUMMARY:
This is a multicenter post-marketing clinical follow-up study to collect safety and performance data in a prospective cohort of patients who will have undergone coil embolization using the ED Coil and ED Detach Generator v4.

ELIGIBILITY:
Inclusion Criteria:

* Patients are over 18 years of age.
* Patients will undergo catheter embolization using the Kaneka ED Coil with the ED Detach Generator v4 for aneurysm, arteriovenous malformation (AVM), or arteriovenous fistula (AFV)
* The patient, or his/her representative, has agreed to the informed consent.

Exclusion Criteria:

* The patient, or his/her representative, is unwilling or unable to agree to the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with an aneurysm, arteriovenous malformation, or arteriovenous fistula and eligible for endovascular treatment with ED Coil and ED Detach Generator v4.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Performance Measure | At 6 months
  The recanalization in aneurysms will be classified using the Raymond-Roy Classification. The outcomes following embolization of arteriovenous malformations and arteriovenous fistula will be classified as follows complete occlusion/subtotal occlusion/ partial occlusion
Performance Measure | At 12 months
  The recanalization in aneurysms will be classified using the Raymond-Roy Classification. The outcomes following embolization of arteriovenous malformations and arteriovenous fistula will be classified as follows complete occlusion/subtotal occlusion/ partial occlusion
Safety Measure - Assessment of Adverse Events | During 12 months
  All adverse events will be recorded, along with their seriousness and relatedness to the device or the procedure.
Technical Measure | At embolization procedure, an average of 1 week
  The technical properties of the ED Electrodetach Generator v4 will be assessed by successful coil detachment (yes/no)
Technical Measure | At embolization procedure, an average of 1 week
  The technical properties of the ED Electrodetach Generator v4 will be assessed by the the number of detachment attempts

CONTACTS AND LOCATIONS:
Locations (3):
- UZA Atwerp, Edegem, Antwerp, Belgium
- Germany (2):
  - Knappschaftskrankenhaus Bochum, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein